CLINICAL TRIAL: NCT06480253
Title: Variation of Cerebral Blood Flow Depending on the Interface Chosen During Continuous Positive Airway Pressure Ventilation
Brief Title: Cerebral Blood Flow: Helmet vs Oronasal Mask During Continuous Positive Airway Pressure Ventilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Roberto Cosentini, Director of Emergency Department, Papa Giovanni XXIII Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CBF - Helmet vs Mask
Record Dates: First submitted 2024-06-13; First posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Ventilation Therapy
Keywords: Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Open Label, randomized, controlled with crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Helmet (Experimental): Partecipants will be started on Continuous Positive Airway Pressure using the Helmet interface
  Interventions: Device: Helmet Continuous Positive Airway Pressure
- Oronasal Mask (Active Comparator): Partecipants will be started on Continuous Positive Airway Pressure using the oronasal mask interface
  Interventions: Device: Oronasal Mask Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Helmet Continuous Positive Airway Pressure — Partecipants will be started on Continuous Positive Airway Pressure at 10 cmH2O on inspired fraction of oxygen (FiO2)= 21% with the Helmet interface for a duration of 5 minutes while laying down on a stretcher with head elevated at 60°
  Arms: Helmet
Device: Oronasal Mask Continuous Positive Airway Pressure — Partecipants will be started on Continuous Positive Airway Pressure at 10 cmH2O on Inspired fraction of oxygen (FiO2)= 21% with the oronasal mask interface for a duration of 5 minutes while laying down on a stretcher with head elevated at 60°
  Arms: Oronasal Mask

SUMMARY:
In this trial the investigators will evaluate blood flow in common carotid artery of healthy subjects treated with Continuous Positive Airway Pressure (CPAP) Ventilation, comparing two different devices: oronasal mask versus Helmet. The hypothesis is that Helmet CPAP reduces carotid flow compared to oronasal mask.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Ability to give informed consent

Exclusion Criteria:

* known cardiac pathologies
* known pulmonary pathologies
* known vascular pathologies
* history of concussion
* history of headache

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Common carotid artery flow | 4 consecutive heart beats at the end of the intervention
  Left common carotid artery flow, expressed as ml/min measured with pulsed wave doppler with ultrasound

SECONDARY OUTCOMES:
Mean arterial blood pressure | single measure, at the end of the intervention
  Non invasive mean arterial blood pressure on left arm
Peripheral vascular resistance | 4 consecutive heart beats at the end of the intervention
  Peripheral vascular resistance measured in left common carotid artery, measured with pulsed wave doppler with ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cosentini, MD, Study Director — Ospedale Papa Giovanni XXIII
Locations (1):
- Ospedale Papa Giovanni XXIII, Bergamo, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD will be given on request for scientific porpoise after the publication of the results of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be given on request for scientific porpoise after the publication of the results of the study
Access Criteria: Data will be shared by email

REFERENCES:
- [Background] Haring HP, Hormann C, Schalow S, Benzer A. Continuous positive airway pressure breathing increases cerebral blood flow velocity in humans. Anesth Analg. 1994 Nov;79(5):883-5. doi: 10.1213/00000539-199411000-00011. PMID 7978404
- [Background] Scala R, Turkington PM, Wanklyn P, Bamford J, Elliott MW. Effects of incremental levels of continuous positive airway pressure on cerebral blood flow velocity in healthy adult humans. Clin Sci (Lond). 2003 Jun;104(6):633-9. doi: 10.1042/CS20020305. PMID 12580765
- [Background] Kolbitsch C, Lorenz IH, Hormann C, Schocke M, Kremser C, Zschiegner F, Felber S, Benzer A. The impact of increased mean airway pressure on contrast-enhanced MRI measurement of regional cerebral blood flow (rCBF), regional cerebral blood volume (rCBV), regional mean transit time (rMTT), and regional cerebrovascular resistance (rCVR) in human volunteers. Hum Brain Mapp. 2000 Nov;11(3):214-22. doi: 10.1002/1097-0193(200011)11:3<214::AID-HBM70>3.0.CO;2-I. PMID 11098799
- [Background] Yiallourou TI, Odier C, Heinzer R, Hirt L, Martin BA, Stergiopulos N, Haba-Rubio J. The effect of continuous positive airway pressure on total cerebral blood flow in healthy awake volunteers. Sleep Breath. 2013 Mar;17(1):289-96. doi: 10.1007/s11325-012-0688-0. Epub 2012 Mar 22. PMID 22434361